CLINICAL TRIAL: NCT00193622
Title: A Phase II Trial of Bevacizumab and Erlotinib in the Treatment of Patients With Carcinoma of Unknown Primary Site
Brief Title: Bevacizumab and Erlotinib in the Treatment of Patients With Carcinoma of Unknown Primary Site
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI UNKPRI 15; AVF 2968s
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Neoplasms, Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Bevacizumab; Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Bevacizumab
Drug: Erlotinib

SUMMARY:
This trial will investigate the combination of bevacizumab, and erlotinib in patients with adenocarcinoma or poorly differentiated carcinoma of unknown primary site. Bevacizumab and erlotinib are relatively well-tolerated and have non-overlapping toxicity profiles. This trial will be one of the first clinical trials to evaluate a combination of targeted agents in the treatment of a solid tumor.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Bevacizumab + Erlotinib

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Carcinoma of unknown primary site confirmed by biopsy
* Measurable disease
* ECOG performance status must be 0-1
* Adequate bone marrow, liver and kidney
* Understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age< 18 years
* May not have received EGFR inhibitors
* History of acute myocardial infarction within 6 months
* Clinically significant cardiovascular disease
* Moderate to severe peripheral vascular disease.
* History of stroke within 6 months
* History of abdominal fistula, perforation, or abscess within 6 months
* Active concurrent infections
* Serious underlying medical conditions
* Active brain metastases
* Women who are pregnant or lactating.
* PEG or G-tube
* Proteinuria
* Any nonhealing wound, ulcer, or bone fracture.
* Any clinical evidence or history of bleeding, clotting or coagulopathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-04; Primary Completion 2005-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Time to progression
Overall survival
Overall tolerability
Overall toxicity

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Farley C, Thompson DS, Shipley DL, Greco FA; Minnie Pearl Cancer Research Network. Phase II trial of bevacizumab and erlotinib in carcinomas of unknown primary site: the Minnie Pearl Cancer Research Network. J Clin Oncol. 2007 May 1;25(13):1747-52. doi: 10.1200/JCO.2006.09.3047. PMID 17470864
- See also: Published article in the Journal of Clinical Oncology — http://jco.ascopubs.org/cgi/content/full/25/13/1747